CLINICAL TRIAL: NCT06704087
Title: Télésurveillance de Patients Porteurs d'Une Plaie Chronique à l'Aide d'Une Solution numérique MyDerm : étude de faisabilité
Brief Title: Telemonitoring of Chronic Wound Patients Using MyDerm, a Digital Solution: Feasibility Study
Acronym: PIXAPROM
Status: Completed | Type: Observational
Sponsor: Pixacare (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024/001/Pixacare
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2024-11

CONDITIONS: Single Chronic Wound; Lower Limb Wound
Keywords: chronic wound; telemonitoring; patient satisfaction; caregivers satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — There is no biospecimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Telemonitoring: patients with chronic wounds of the lower limb benefiting from the digital solution for remote monitoring of healing.

SUMMARY:
The aim of this study is to assess the feasibility of integrating myDerm for remote monitoring of chronic wounds into everyday practice, for patients over 18 years of age suffering from a single chronic wound of the lower limb (more than 6 weeks old).

Outcome measure 1 :

Evaluate patient satisfaction after 2 months of using the MyDerm solution.

Outcome measure 2 :

1. Evaluate caregiver satisfaction after 2 months of patient use of MyDerm solution.
2. Assess patient use (compliance, frequency) of MyDerm solution
3. Evaluate caregiver use of PIXACARE solution
4. Evaluate the impact of patients' socio-demographic characteristics (age, gender, level of education: primary/secondary/tertiary, rural/urban) on use of the MyDerm solution.
5. Evaluate the impact of patients' clinical characteristics on the use of the MyDerm solution.

Researchers will compare standard of care arm vs remote monitoring arm.

As part of remote monitoring, patients are invited to take photos of their wounds using their smartphone, and to answer a simple questionnaire to look for signs of complications. To assess satisfaction, the patient will complete a questionnaire after 2 months' use, using a 7-level Likert scale.

DETAILED DESCRIPTION:
Observational, monocentric study of patients with chronic wounds of the lower limb benefiting from the digital solution for remote monitoring of wound healing.

Clinical data will be collected by the investigating team during the primary consultation.

Patient satisfaction surveys will be sent in paper format to patients at the consultation scheduled at the end of the two-month follow-up period.

Caregiver" satisfaction surveys will be sent in paper format to caregivers at the end of the study.

The number of actions taken in response to an alert (by telephone, by message, organization of a physical consultation, organization of a teleconsultation, hospitalization) will be recorded in the post-alert action traceability form

ELIGIBILITY:
Inclusion Criteria:

* Patient with a single chronic wound of the lower limb (more than 6 weeks)
* Benefiting from the MyDerm digital wound-healing monitoring solution
* Patient aged 18 or over
* Informed patient who has not objected to the use of data

Exclusion Criteria:

* Patient refusing to participate in the study
* Patient included in a clinical trial
* Patient with a life expectancy shorter than the duration of the study
* Patient with cognitive impairment
* Inability to install or use the medical device for technical reasons (lack of internet connection, lack of 4G coverage or more, lack of smartphone)
* Patient requiring home hospital care
* Patient requiring Follow-up and rehabilitation care
* Pregnant or breast-feeding women
* Patient with a previously infected wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic wounds of the lower limb benefiting from the digital solution for remote monitoring of healing at hospital
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Response to questionnaire completed after two months of use | At 2 months
  The satisfaction questionnaire using a 7-point Likert scale

SECONDARY OUTCOMES:
Responses to the caregiver questionnaire completed at the end of the study using a 7-point Likert scale | At 2 months
  The satisfaction questionnaire using a 7-point Likert scale
Patient use of the MyDerm solution | At 2 months
  A. Number of patients with at least one telefile B. Total number of teledeposits generated per patient during the follow-up period C. Number of teledeposits per week per patient over the entire follow-up period (evolution of usage over the follow-up period)
The impact of patients' socio-demographic characteristics on use of the MyDerm solution | At 2 months
  Number of patients with at least one telefile
The impact of patients' socio-demographic characteristics on use of the MyDerm solution | AT 2 months
  Total number of teledeposits generated per patient during follow-up period
The impact of patients' socio-demographic characteristics on use of the MyDerm solution | AT 2 months
  Number of teledeposits per week per patient over the entire follow-up period (evolution of usage over the follow-up period)
Use of PIXACARE solution by caregivers | At 2 months
  Number of telemonitoring records opened per patient by the medical team during the follow-up period.
Use of PIXACARE solution by caregivers | AT 2 months
  Total number of alerts and number of alerts per patient during follow-up period
Use of PIXACARE solution by caregivers | At 2 months
  Number of actions by telephone related to an alert
Use of PIXACARE solution by caregivers | At 2 months
  Number of e-mail related to an alert
Use of PIXACARE solution by caregivers | AT 2 months
  Number of organization of a physical consultation related to an alert
Use of PIXACARE solution by caregivers | At 2 months
  Number of organization of a teleconsultation
Use of PIXACARE solution by caregivers | At 2 months
  Number of hospitalization related to an alert

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France, France